CLINICAL TRIAL: NCT01267682
Title: Reserve For Delirium Superimposed On Dementia (DSD)
Brief Title: Cognitive Intervention For Delirium in Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Ann Kolanowski, Professor of Nursing, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR012242 (NIH)
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Delirium; Dementia
Keywords: Delirium; Dementia; Non-pharmacological Intervention; Post-acute care
MeSH Terms: conditions — Delirium; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Participants receive standard clinical care
- Treatment (Experimental): Behavioral: cognitive stimulation
  Interventions: Behavioral: Cognitive Stimulation

INTERVENTIONS:
Behavioral: Cognitive Stimulation — Thirty minutes of cognitive stimulation delivered daily for thirty minutes.
  Arms: Treatment

SUMMARY:
The purpose of this study is to test the effectiveness of cognitively stimulating activities for resolving delirium in people with dementia.

DETAILED DESCRIPTION:
The primary aim in this RCT is to test the efficacy of Recreational Stimulation for Elders as a Vehicle to resolve DSD (RESERVE- DSD). The investigators will randomize 256 subjects, newly admitted to post acute care, to intervention (RESERVE-DSD) or control (usual care). Intervention subjects will receive 30-minute sessions of tailored cognitively stimulating recreational activities for up to 30 days. The investigators hypothesize that subjects who receive RESERVE-DSD will have: decreased severity and duration of delirium; greater gains in attention, orientation, memory, abstract thinking, and executive functioning; and greater gains in physical function compared to subjects with DSD who receive usual care. The investigators will also evaluate potential moderators of intervention efficacy (lifetime of complex mental activities and APOE status). The secondary aim is to describe the costs associated with RESERVE-DSD.

ELIGIBILITY:
Inclusion Criteria:

* presence of delirium
* mild to moderate cognitive impairments
* 65 years of age or older
* English speaking
* community-dwelling
* legally authorized representative available

Exclusion Criteria:

* severe vision or hearing problems
* diagnosis of

  1. major depression
  2. Parkinson's with Lewy Body disease
  3. Huntington's disease
  4. normal pressure hydrocephalus
  5. seizure disorder
  6. subdural hematoma
  7. head trauma
  8. known structural brain abnormalities
  9. acute CVA/stroke
  10. acute psychiatric condition
* life expectancy < 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 283 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Confusion Assessment Method | Averaged over 30 days or until discharge, whichever comes first
Delirium Rating Scale | Averaged over 30 days or until discharge, whichever comes first

SECONDARY OUTCOMES:
Attention | Averaged over 30 days or until discharge, whichever comes first
Memory | Averaged over 30 days or until discharge, whichever comes first
Abstract Thinking | Averaged over 30 days or until discharge, whichever comes first
Orientation | Averaged over 30 days or until discharge, whichever comes first
Executive Function | Averaged over 30 days or until discharge, whichever comes first
Physical Function | Averaged over 30 days or until discharge, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Kolanowski, PhD, RN, Principal Investigator — Penn State University; Donna M Fick, PhD, RN, Principal Investigator — Penn State University
Locations (9):
- United States (9):
  - Centre Crest Nursing Home, Bellefonte, Pennsylvania
  - The Meadows Manor, Dallas, Pennsylvania
  - Spring Creek Rehabilitation and Nursing Center, Harrisburg, Pennsylvania
  - Windy Hill Village, Philipsburg, Pennsylvania
  - Mountain View, Scranton, Pennsylvania
  - Brookline Nursing & Rehabilitation Center, State College, Pennsylvania
  - Hearthside Nursing and Rehabilitation Center, State College, Pennsylvania
  - Hearthside Nursing Home, State College, Pennsylvania
  - The Village at Penn State, State College, Pennsylvania

REFERENCES:
- [Background] Yevchak A, Steis M, Diehl T, Hill N, Kolanowski A, Fick D. Managing delirium in the acute care setting: a pilot focus group study. Int J Older People Nurs. 2012 Jun;7(2):152-62. doi: 10.1111/j.1748-3743.2012.00324.x. Epub 2012 Apr 18. PMID 22513181
- [Background] Kolanowski AM, Fick DM, Litaker MS, Clare L, Leslie D, Boustani M. Study protocol for the recreational stimulation for elders as a vehicle to resolve delirium superimposed on dementia (Reserve For DSD) trial. Trials. 2011 May 11;12:119. doi: 10.1186/1745-6215-12-119. PMID 21569370
- [Background] Kolanowski AM, Fick DM, Clare L, Steis M, Boustani M, Litaker M. Pilot study of a nonpharmacological intervention for delirium superimposed on dementia. Res Gerontol Nurs. 2011 Jul;4(3):161-7. doi: 10.3928/19404921-20101001-98. Epub 2010 Oct 29. PMID 21053841
- [Background] Kolanowski AM, Fick DM, Clare L, Therrien B, Gill DJ. An intervention for delirium superimposed on dementia based on cognitive reserve theory. Aging Ment Health. 2010 Mar;14(2):232-42. doi: 10.1080/13607860903167853. PMID 20336555
- [Background] Hill NL, Kolanowski AM, Gill DJ. Plasticity in Early Alzheimer's Disease: An Opportunity for Intervention. Top Geriatr Rehabil. 2011 Oct;27(4):257-267. doi: 10.1097/tgr.0b013e31821e588e. PMID 22904596
- [Background] Kolanowski AM, Fick DM, Yevchak AM, Hill NL, Mulhall PM, McDowell JA. Pay attention! The critical importance of assessing attention in older adults with dementia. J Gerontol Nurs. 2012 Nov;38(11):23-7. doi: 10.3928/00989134-20121003-05. Epub 2012 Oct 15. PMID 23066682
- [Background] Kolanowski A, Bossen A, Hill N, Guzman-Velez E, Litaker M. Factors associated with sustained attention during an activity intervention in persons with dementia. Dement Geriatr Cogn Disord. 2012;33(4):233-9. doi: 10.1159/000338604. Epub 2012 May 31. PMID 22652933
- [Background] Kolanowski A, Mulhall P, Yevchak A, Hill N, Fick D. The triple challenge of recruiting older adults with dementia and high medical acuity in skilled nursing facilities. J Nurs Scholarsh. 2013 Dec;45(4):397-404. doi: 10.1111/jnu.12042. Epub 2013 Jul 16. PMID 23859475
- [Background] Yevchak AM, Fick DM, McDowell J, Monroe T, May K, Grove L, Kolanowski AM, Waller JL, Inouye SK. Barriers and facilitators to implementing delirium rounds in a clinical trial across three diverse hospital settings. Clin Nurs Res. 2014 Apr;23(2):201-15. doi: 10.1177/1054773813505321. Epub 2013 Oct 11. PMID 24121464
- [Result] Kolanowski AM, Hill NL, Kurum E, Fick DM, Yevchak AM, Mulhall P, Clare L, Valenzuela M. Gender differences in factors associated with delirium severity in older adults with dementia. Arch Psychiatr Nurs. 2014 Jun;28(3):187-92. doi: 10.1016/j.apnu.2014.01.004. Epub 2014 Feb 5. PMID 24856271
- [Result] Hill NL, Kolanowski AM, Fick D, Chinchilli VM, Jablonski RA. Personality as a moderator of cognitive stimulation in older adults at high risk for cognitive decline. Res Gerontol Nurs. 2014 Jul-Aug;7(4):159-70. doi: 10.3928/19404921-20140311-01. Epub 2014 Mar 18. PMID 24635006